CLINICAL TRIAL: NCT01447043
Title: AURA Study: A Retrospective Non-interventional Study (NIS) to Assess the Effectiveness of Existing Anti vascUlar Endothelial Growth Factor (Anti VEGF) Treatment Regimens in Patients With Wet Age-related Macular Degeneration (wAMD)
Brief Title: Study to Assess the Effectiveness of Existing Anti vascUlar Endothelial Growth Factor (Anti VEGF) in Patients With Wet Age-related Macular Degeneration (wAMD) (AURA)
Acronym: AURA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15913; NN1101 (Other: company internal)
Record Dates: First submitted 2011-09-20; First posted 2011-10-05 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Ophthalmology, Macular Degeneration
Keywords: retrospective studies
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Patients with wet AMD treated with ranibizumab as prescribed by physician

SUMMARY:
Retrospective, non-interventional, observational multi-center field study. Patients diagnosed with wet Age-related macular degeneration (wAMD) and having started treatment with ranibizumab between January 1, 2009 and August 31, 2009 must be consecutively screened and, if eligible, enrolled. Patients will be followed up at maximum until August 31, 2011. Switch to any other Anti vascUlar endothelial growth factor (anti VEGF) treatment will be documented and followed up. For each patient, demographics, medical history, administered treatments, results of ocular and visual assessments and other tests (where available) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of wet age-related macular degeneration
* Start of Anti vascUlar endothelial growth factor (anti VEGF) therapy with ranibizumab between January 1, 2009 and August 31, 2009
* Informed consent form signed, where required

Exclusion Criteria:

* Participation in an investigational study during anti-VEGF therapy (from start up to August 31, 2011) that involved treatment with any drug or medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been diagnosed to suffer from wet AMD and must have started anti-VEGF treatment with ranibizumab between January 1, 2009, and August 31, 2009.
Sampling Method: Non-Probability Sample
Enrollment: 2609 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity after start of Anti vascUlar endothelial growth factor (anti VEGF) therapy with ranibizumab, assessed by Early Treatment Diabetic Retinopathy (ETDRS) or Snellen chard | Baseline and 24 months

SECONDARY OUTCOMES:
Demographic characteristics of patients included in the study (Age, Sex, Race) | Baseline
Mean time from first clinical presentation to diagnosis | Time from first clinical presentation to diagnosis: Up to 36 months
Mean time from diagnosis to treatment | Time from diagnosis to treatment: Up to 24 months
Mean time from diagnosis to end of follow-up | Time from diagnosis to end of follow-up: 48 months
Mean change of visual acuity, from diagnosis to end of follow-up, assessed by Early Treatment Diabetic Retinopathy (ETDRS) or SNELLEN | Baseline and 24 months
Mean change of retinal thickness from diagnosis to end of follow-up, assessed by Optical Coherence Tomography (OCT) | Baseline and 24 months
Mean change of lesion size from diagnosis to end of follow-up, assessed by Fluorescein Angiography (FA) | Baseline and 24 months
Average number of treatments given from diagnosis to end of follow-up | After 24 months
Vital Signs (blood pressure, heart rate, temperature) of patients included in the study | Baseline
Medical and surgical history (diseases and surgeries) of patients included in the study | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Many Locations, Australia
- Many Locations, Canada
- Many Locations, France
- Many Locations, Germany
- Many Locations, Ireland
- Many Locations, Italy
- Many Locations, Japan
- Many Locations, Netherlands
- Many Locations, United Kingdom
- Many Locations, Venezuela

REFERENCES:
- [Derived] Holz FG, Tadayoni R, Beatty S, Berger A, Cereda MG, Hykin P, Staurenghi G, Wittrup-Jensen K, Altemark A, Nilsson J, Kim K, Sivaprasad S. Key drivers of visual acuity gains in neovascular age-related macular degeneration in real life: findings from the AURA study. Br J Ophthalmol. 2016 Dec;100(12):1623-1628. doi: 10.1136/bjophthalmol-2015-308166. Epub 2016 Mar 30. PMID 27030279
- [Derived] Holz FG, Tadayoni R, Beatty S, Berger A, Cereda MG, Cortez R, Hoyng CB, Hykin P, Staurenghi G, Heldner S, Bogumil T, Heah T, Sivaprasad S. Multi-country real-life experience of anti-vascular endothelial growth factor therapy for wet age-related macular degeneration. Br J Ophthalmol. 2015 Feb;99(2):220-6. doi: 10.1136/bjophthalmol-2014-305327. Epub 2014 Sep 5. PMID 25193672